CLINICAL TRIAL: NCT01465477
Title: Influenza Vaccination in Patients Suffering From Fibromyalgia
Brief Title: Influenza Vaccination in Fibromyalgia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0332-11-TLV; 0332-11-TLV (Registry Identifier: Tel Aviv Medical Center IRB)
Record Dates: First submitted 2011-10-24; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-10

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia; Influenza vaccination
MeSH Terms: conditions — Fibromyalgia; Influenza, Human

ARMS (2):
- Fibromyalgia arm (Experimental): Patients fulfilling ACR 1990 Criteria for classification of Fibromyalgia, receiving the vaccination.
  Interventions: Biological: Inactivated split virion Influenza vaccine
- Heathy controls (Experimental): Healthy controls receiving Influenza vaccination
  Interventions: Biological: WHO recommended 2011 Influenza vacccine

INTERVENTIONS:
Biological: Inactivated split virion Influenza vaccine — WHO recommended 2011 Influenza vaccine
  Arms: Fibromyalgia arm
Biological: WHO recommended 2011 Influenza vacccine — WHO recommended 2011 Influenza vacccine
  Arms: Heathy controls

SUMMARY:
Fibromyalgia is a clinical syndrome characterized by the presence of chronic widespread pain accompanied by tenderness and fatigue. Central sensitization is considered to be a major pathogenetic feature of fibromyalgia. While the etiology of fibromyalgia is incompletely understood, it is generally considered to result from the interaction between an appropriate genetic background and the exposure of a susceptible individual to various inciting "triggers". These have included among others physical trauma, infection, stress etc.

The possible role of vaccination in causing or exacerbating fibromyalgia has been previously raised. Thus, gulf war syndrome, an entity with considerable clinical overlap with fibromyalgia, has been considered to have a possible link with the exposure to multiple vaccinations. More recently a theory has been advanced regarding the possibility that vaccination - related adjuvants may induce a multisystem disorder characterized by symptoms such as fatigue, cognitive impairment and arthralgia (the so called ASIA syndrome).

The investigators have previously established the safety and efficacy of influenza vaccination in Rheumatoid arthritis patients.

In view of this background it is of considerable clinical importance to ascertain both the efficacy and safety of vaccination in patients suffering from fibromyalgia.

DETAILED DESCRIPTION:
Fifty patients with fibromyalgia and 30 healthy, age - matched controls will participate in the study.

The classification of fibromyalgia will be performed by applying the 1990 ACR criteria.

After signing informed consent, all subjects will be vaccinated with the inactivated split virion vaccine, recommended by the WHO this fall.

Patients will be evaluated at weeks 0 and 6 weeks later. Clinical evaluation will be based on the Fibromyalgia Impact Questionnaire and the 2010 Fibromyalgia Severity Scale.

ESR and CRP Blood will be collected on the day of vaccination and 6 weeks later.

The immunogenicity of the vaccine will be tested by Haemagglutination inhibition (HI) test.

Influenza virus has two important surface glycoproteins: the haemagglutinin (HA) and the neuraminidase (NA). Antigenic classification and subtyping of influenza viruses is based on these two glycoproteins. HA plays a key role in virus cell entry by binding to cell surface receptors, which are found also on red blood cells of certain species. Binding to red cells results in haemagglutination, which can be observed as a carpet of agglutinated red cells at the bottom of a tube or microtitre well. In the HI test, antibody directed against the viral haemagglutinins block the virus from binding to the blood cells and thus inhibits the haemagglutination reaction.

The pre- and post immunization HI antibodies were tested at the Central Virology Laboratory of the Israeli Ministry of Health using the HI test according to a standard WHO procedure 16. Sera will be separated, code labeled, and stored at -20°C until tested. Sera will be treated with receptor destroying enzyme cholera filtrate to remove non-specific inhibitors, and with Turkey red blood cells to remove non-specific agglutinins. The treated sera will be tested by HI test against the three antigens included in the vaccine: A/California (CAL), A/Wisconsin and B/Malaysia. The working dilution (test dose) of each antigen contained four haemagglutinin units in 25 µl of antigen. Test doses will be diluted in phosphate buffered saline (PBS) and added to serial dilution of antiserum. The haemagglutinin inhibition titer will be determined as the highest dilution of serum that completely inhibits haemagglutination of red blood cells.

The titer of an antiserum not showing any inhibition will be recorded as <10. Humoral response will be defined as either a fourfold or more rise in titer, or a rise from a non-protective baseline level of <1/40 to 1/40 in HI antibodies four weeks after vaccination 17,18. Geometric mean titers of antibody will be calculated to assess the immunity of the whole group.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 year old age
* Capable to sign a informed consent
* Suffering from fibromyalgia (ACR criteria)

Exclusion Criteria:

* Known allergy to influenza vaccine
* Allergy to eggs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
proportion of patients who achieve a titer of antibodies above 1/40, against each of the antigens included in the vaccine | Six weeks

SECONDARY OUTCOMES:
Number of adverse events | Six weeks
  The occurrence of vaccine - related adverse events (allergic reactions, pain at injection site, fever etc) will be documented.
Clinical changes post - vaccination | Six weeks
  Clinical evaluation of Fibromyalgia patients will be performed on follow up, including a tender point count and documentation of the Fibromyalgia severity scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob N Ablin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Rheumatology Institute, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Elkayam O, Amir S, Mendelson E, Schwaber M, Grotto I, Wollman J, Arad U, Brill A, Paran D, Levartovsky D, Wigler I, Caspi D, Mandelboim M. Efficacy and safety of vaccination against pandemic 2009 influenza A (H1N1) virus among patients with rheumatic diseases. Arthritis Care Res (Hoboken). 2011 Jul;63(7):1062-7. doi: 10.1002/acr.20465. PMID 21425247
- [Background] Ablin JN, Shoenfeld Y, Buskila D. Fibromyalgia, infection and vaccination: two more parts in the etiological puzzle. J Autoimmun. 2006 Nov;27(3):145-52. doi: 10.1016/j.jaut.2006.09.004. Epub 2006 Oct 30. PMID 17071055
- [Background] Meroni PL. Autoimmune or auto-inflammatory syndrome induced by adjuvants (ASIA): old truths and a new syndrome? J Autoimmun. 2011 Feb;36(1):1-3. doi: 10.1016/j.jaut.2010.10.004. Epub 2010 Nov 3. PMID 21051205